CLINICAL TRIAL: NCT03672149
Title: A Prospective, Open-Label Study of the Safety and Therapeutic Drug Monitoring of Continuous Infusion Cefazolin Through the Addition of the Cefazolin Into the Continuous Renal Replacement Therapy Solution.
Brief Title: Safety and Therapeutic Drug Monitoring of Cefazolin in Continuous Renal Replacement Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Collaborators: The Center for Pediatric Pharmacotherapy (Unknown)
Responsible Party: Principal Investigator, Jeffrey J. Cies,PharmD,MPH,BCPS-AQ ID,BCPPS,FCCP,FCCM,FPPAG, Principal Investigator, Drexel University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1805006375
Record Dates: First submitted 2018-09-10; First posted 2018-09-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Renal Replacement Therapy; Pharmacokinetics
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: 1. If cefazolin is part of the empiric or definitive treatment regimen, it will be mixed in the CRRT solution(s) and administered via a continuous infusion to obtain treatment, pharmacokinetic, and safety data .
  2. If cefazolin is not part of the empiric or definitive treatment regimen, it will be mixed in the CRRT solution(s) and administered via a continuous infusion to obtain pharmacokinetic, and safety data .
  3. If a patient does not require any anti-microbial therapy, cefazolin will be given via the CRRT solution(s) to solely obtain pharmacokinetic and safety data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Infection needing cefazolin (Other): a) If a patient requires antimicrobial therapy for a proven or suspected infection at the time of CRRT initiation or at any time receiving CRRT, they are eligible for inclusion. If cefazolin is part of the empiric or definitive treatment regimen, it will be mixed in the CRRT solution(s) and administered via a continuous infusion to obtain pharmacokinetic and safety data of administering cefazolin via the CRRT solution and infection treatment related data. For this indication, pharmacokinetic and safety data will be obtained for the duration the patient receives cefazolin via the CRRT solution(s) for the proven or suspected infection as dictated by the primary team caring for the patient.
  Interventions: Drug: Cefazolin
- Infection not needing cefazolin (Other): b) If a patient is deemed a candidate for CRRT and requires therapy with any anti-microbial for a proven or suspected infection not requiring cefazolin as part of the anti-microbial drug regimen, administration of cefazolin via the CRRT solution(s) will occur to solely obtain pharmacokinetic and safety data. For this indication, pharmacokinetic and safety data will be obtained for a 72-96-hour duration.
  Interventions: Drug: Cefazolin
- No infection (Other): c) If a patient is deemed a candidate for CRRT and does not require any anti-microbial therapy, administration of cefazolin via the CRRT solution(s) will occur to solely obtain pharmacokinetic and safety data. For this indication, pharmacokinetic and safety data will be obtained for a 72-96-hour duration.
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — Mixing cefazolin into the CRRT solution(s) for delivery as a continuous infusion
  Other Names: CRRT solutions

SUMMARY:
This investigation is intended to collect safety information for the technique of mixing cefazolin in the CRRT solution on the CRRT circuit, the patient, in addition to collecting information regarding the ability to obtain therapeutic cefazolin serum concentrations

DETAILED DESCRIPTION:
This investigation is intended to collect safety information for the technique of mixing cefazolin in the CRRT solution on the CRRT circuit, the patient, in addition to collecting information regarding the ability to obtain therapeutic cefazolin serum concentrations in addition to utilizing a dosing algorithm to adjust the cefazolin concentration in the CRRT solution.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible to participate in the study must have a need for continuous renal replacement therapy (CRRT) of any modality:

1. CVVH-continuous veno-venous hemofiltration
2. CVVHD-continuous veno-venous hemodialysis
3. CVVHDF-continuous veno-venous hemodiafiltration

Exclusion Criteria:

Patients will be considered ineligible if they meet any of the following criteria:

1. History of any moderate or severe hypersensitivity or allergic reaction to cefazolin (a history of mild rash followed by uneventful re-exposure and/or red man syndrome is not a contraindication)
2. Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator)
3. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data
4. Females that are pregnant or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cefazolin serum levels | 72-96 hours
  Therapeutic serum cefazolin levels. Serum samples will be obtained at specified intervals during the course of CRRT for cefazolin concentration determination.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Christopher's Hospital for Children, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No